CLINICAL TRIAL: NCT03936478
Title: A Phase II Study of Real-Time MRI-Guided 3-Fraction Accelerated Partial Breast Irradiation in Early Breast Cancer (MAPBI)
Brief Title: Real-Time MRI-Guided 3-Fraction Accelerated Partial Breast Irradiation in Early Breast Cancer
Acronym: MAPBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW18099; 2019-0322 (Other: Institutional Review Board); SMPH\HUMAN ONCO\HUMAN ONCO (Other: UW Madison); A533300 (Other: UW Madison); NCI-2019-03111 (Registry Identifier: NCI Trial ID); Protocol Version 5/10/2021 (Other: UW Madison)
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; DCIS; LCIS
Keywords: cosmesis; cosmetic; breast-conserving therapy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Intervention Model Description: This study will have a lead-in phase consisting of 10 patients, followed for 6-months from the date of completion of radiotherapy for the tenth patient. The second phase of accrual (20 patients) will commence only if three or fewer patients (3/10=30%) have CTCAE v 5.0 grade 3 or higher skin toxicity (radiation dermatitis) or Lövey et al. grade 3 or higher fat necrosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 8.2 Gy Radiation Therapy (Experimental): Accelerated partial breast irradiation using 3 x 8.2 Gy to the lumpectomy cavity with a 3mm PTV margin. Treatment duration will be 5-6 days and treatments will be on alternative weekdays, with a minimum interval of 40 hours between subsequent fractions.
  Interventions: Radiation: MRIdian Radiation Treatment Unit

INTERVENTIONS:
Radiation: MRIdian Radiation Treatment Unit — partial breast irradiation using 3 x 8.2 Gy to the lumpectomy cavity with a 3mm planning tumor volume (PTV) margin

SUMMARY:
This trial will investigate a novel 3-fraction radiation regimen for participants undergoing breast-conserving therapy (BCT) for early breast cancer that will: 1) significantly reduce the duration of treatment and can be completed in one-week (5 working days) and 2) MRI-guided radiotherapy (MRIdian) would limit the volume of normal tissue radiated and therefore resultant toxicity. The hypothesis is that 3-fraction radiation therapy can be delivered safely without compromising the therapeutic ratio. Participants can expect to be on study for follow up up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

For all participants

* Participants should have no contraindications to undergo MRI scan as part of radiotherapy planning and treatment.
* Lumpectomy cavity must be clearly visible on CT and MRI scan at radiotherapy simulation.
* Pregnancy test negative in women of child bearing potential (WOCBP).
* The participant must consent to be in the study and must have signed an approved consent form conforming with institutional guidelines.
* Participants with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior and are deemed by their physician to be at low risk for recurrence. Participants with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

For participants with Invasive Carcinoma

* Suitable:

  * Age: >=50 years

    * Margins: Negative by at least 2 mm
    * T Stage: Tis or T1
* Cautionary:

  * Age: 40-49 years

    * Margins: Negative by at least 2 mm
    * T Stage: Tis or T1 OR
  * Age: >=50 years IF participant has at least 1 of the pathologic factors below and does not have any "unsuitable" factors (below)

    * Pathologic Factors:

      * Size 2.1-3.0 cm (size of the invasive component)
      * T2
      * Close margins (<2 mm)
      * Limited/focal Lymphovascular Space Invasion (LVSI)
      * ER (-)
      * Clinically unifocal with total size 2.1-3.0 cm (Microscopic multifocality allowed, provided the lesion is clinically unifocal (a single discrete lesion by physical examination and ultrasonography/mammography) and the total lesion size (including foci of multifocality and intervening normal breast parenchyma) falls between 2.1 and 3.0 cm).
      * Invasive lobular histology
      * Extensive Intraductal Component (EIC) <=3 cm

For participants with DCIS

* Suitable Criteria, DCIS allowed if all of the following are met:

  * Screen-detected
  * Low to intermediate nuclear grade
  * Size <=2.5 cm
  * Resected with margins negative at >=3mm OR
* Cautionary Criteria:

  * Pure DCIS <=3 cm if "suitable" criteria not fully met

Exclusion Criteria (unsuitable criteria) :

* Men are not eligible for this study.
* BRCA1/2 mutation positivity.
* Age < 40 years (American Society for Radiation Oncology (ASTRO) Unsuitable Criteria).
* Positive resection margins on post operative pathology(ASTRO Unsuitable Criteria).
* Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
* Suspicious micro calcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma (invasive cancer or DCIS) (ASTRO Unsuitable Criteria).
* Pure DCIS >3 cm in size (ASTRO Unsuitable Criteria).
* Presence of extensive intraductal component >30mm (ASTRO Unsuitable Criteria).
* Paget's disease of the nipple.
* History of previous invasive breast cancer, DCIS, synchronous bilateral invasive or non-invasive breast cancer. (Participants with a history of LCIS treated by surgery alone are eligible.)
* Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation.
* Concurrent therapy with any hormonal agents such as raloxifene (Evista®), tamoxifen, Aromatase Inhibitors or other selective estrogen receptor modulators (SERMs), either for osteoporosis or breast cancer prevention or neoadjuvant therapy.
* Breast implants.
* Prior breast or thoracic radiotherapy for any condition or treatment plan that includes regional nodal irradiation.
* Collagen vascular disease, specifically dermatomyositis with a creatinine phosphokinase level above normal or with an active skin rash, systemic lupus erythematosus, or scleroderma.
* Pregnancy or lactation at the time of treatment. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the participant from meeting the study requirements.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Physician Reported Cosmesis: 1-year | up to 1-year
  The Harvard Cosmesis Scale will be used to report cosmesis at 1 year post treatment. The physician will report how the breast looks relative to original appearance or untreated breast (excellent, good, fair, poor). The physician answers 9 questions on a scale of 0-2 where 0 is none, 1 is present but does not affect cosmesis, 2 is present and affects cosmesis. Scoring is objective with lower scores indicating improved conditions.

SECONDARY OUTCOMES:
Participant Quality of Life: BCTOS Survey | up to 5 years
  Participant Quality of Life will be assessed prior to starting treatment, at end of radiotherapy (RT), 4 weeks post RT, 6 months post RT, 12 months post RT and yearly through 5 years by collecting measures from three scales.The Breast Cancer Treatment Outcomes Scale (BCTOS) is a 22-item scale scored 1-4 where 1 is none, 2 is slight, 3 is moderate, and 4 is large. Total score ranges from 22-88 where lower scores indicated better outcomes.
Participant Quality of Life: Convenience of Care Scale | up to 5 years
  Participant Quality of Life will be assessed prior to starting treatment, at end of radiotherapy (RT), 4 weeks post RT, 6 months post RT, 12 months post RT and yearly through 5 years by collecting measures from three scales. The Convenience of Care scale is an 8-item scale scored 0 (not at all) to 10 (a lot). The total score ranges from 0-80 where lower scores indicate less disruptive interventions.
Participant Quality of Life: MOS SF-36 Survey | up to 5 years
  Participant Quality of Life will be assessed prior to starting treatment, at end of radiotherapy (RT), 4 weeks post RT, 6 months post RT, 12 months post RT and yearly through 5 years by collecting measures from three scales.The Medical Outcomes Study Short Form - 36 (MOS SF-36) Vitality scale measures how a participant has felt in the last 4 weeks. 4-items are scored from 1-5 where 1 is all of the time and 5 is none of the time. 4-items are scored from 0 (no pain) to 10 (pain as bad as you can imagine). Total score ranges from 4-60 where lower scores indicate increased vitality.
Physician Reported Cosmesis: 3-year | up to 3 years
  The Harvard Cosmesis Scale will be used to report cosmesis at 1 year post treatment. The physician will report how the breast looks relative to original appearance or untreated breast (excellent, good, fair, poor). The physician answers 9 questions on a scale of 0-2 where 0 is none, 1 is present but does not affect cosmesis, 2 is present and affects cosmesis. Scoring is objective with lower scores indicating improved conditions.
Physician Evaluated Fat Necrosis | up to 5 years
  Fat necrosis will be assessed prior to treatment, at 6 months post RT, at 12 months post RT, and yearly through 5 years, graded as follows: Grade 0 is no fat necrosis, Grade 1 is Asymptomatic fat necrosis (only radiologic and/or cytologic findings), Grade 2 is Symptomatic fat necrosis not requiring medication (palpable mass with or without mild pain), Grade 3 is Symptomatic fat necrosis requiring medication (palpable mass with significant pain), Grade 4 is Symptomatic fat necrosis requiring surgical intervention.
Acute Radiation Toxicity | up to 90 days from completion of radiation therapy
  The NCI's Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 will be used to identify the type and to grade the severity of acute toxicities. Acute toxicities will be scored from the start of radiation to 90 days after completion of radiotherapy and late toxicities will be scored > 90 days from completion of radiation therapy.
Late Radiation Toxicity | up to 5 years
  The NCI's Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 will be used to identify the type and to grade the severity of late toxicities.
Ipsilateral Breast Tumor Recurrence (IBTR) | up to 5 years
  Defined as evidence of invasive or in situ breast cancer (except LCIS) in the ipsilateral breast. Participants who develop clinical evidence of tumor recurrence in the remainder of the ipsilateral breast must have a biopsy of the suspicious lesion to confirm the diagnosis with documentation of the location.
Ipsilateral Regional Nodal Recurrence | up to 5 years
  Defined as the development of tumor in the ipsilateral internal mammary, ipsilateral supraclavicular, ipsilateral infraclavicular and/or ipsilateral axillary nodes, as well as the soft tissue of the ipsilateral axilla, after operation.
Disease Free Survival (DFS) | up to 5 years
  Disease free survival (DFS) defined as the time from start of radiation to the time of documented recurrent disease in the ipsilateral breast or regional nodes (supraclavicular, axillary or internal mammary) or distant sites (e.g. bone, liver, lung or brain).
Overall Survival (OS) | up to 5 years
  Overall survival (OS) defined as the time from start of radiation to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Anderson, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No